CLINICAL TRIAL: NCT00403793
Title: A Phase II -b, Placebo-Controlled Trial Investigating the Efficacy, Safety and Pharmacokinetics of a Subcutaneous Etonogestrel Implant Combined With i.m. Testosterone Undecanoate for Male Contraception
Brief Title: Hormonal Contraception in Healthy Young Men (P42306)(COMPLETED)(P06057)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P06057
Record Dates: First submitted 2006-11-22; First posted 2006-11-27 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Contraception
MeSH Terms: interventions — etonogestrel; testosterone undecanoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): etonogestrel with testosterone undecanoate
  Interventions: Drug: etonogestrel with testosterone undecanoate
- Arm 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: etonogestrel with testosterone undecanoate — 42 or 44 weeks with etonogestrel implant and testosterone undecanoate injections every 10 to 12 weeks
  Arms: Arm 1
Drug: Placebo — 42 or 44 weeks with placebo implant and placebo injections
  Arms: Arm 2

SUMMARY:
Male volunteers receive a new hormonal contraceptive consisting of an implant releasing a hormone and hormone injections in order to investigate the suppressive effect on sperm production and reversibility of sperm production after end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Mentally and physically healthy
* BMI between 18 and 32 kg/m^2
* Two pre-treatment semen samples > 20 million/ml with normal morphology and motility

Exclusion Criteria:

* History or presence of psychiatric disease, liver disease, renal disease, diabetes, cardiovascular disease, any malignancy, prostatic disease, or genitourinary infection
* PSA > 2.5 ng/ml
* Use of drugs known to interfere with pharmacokinetics of steroids
* Use of lipid-lowering drugs

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 350 (Actual)
Dates: Start 2003-10; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
% of men who had a sperm concentration of 1 million/ml or less at week 16. | Week 16

SECONDARY OUTCOMES:
Semen Parameters | At several timepoints during treatment
Reversibility of Suppression | Post-Treatment
Hormones | At several timepoints
Pharmacokinetics | At several timepoints
Safety | At several timepoints

REFERENCES:
- [Result] Mommers E, Kersemaekers WM, Elliesen J, Kepers M, Apter D, Behre HM, Beynon J, Bouloux PM, Costantino A, Gerbershagen HP, Gronlund L, Heger-Mahn D, Huhtaniemi I, Koldewijn EL, Lange C, Lindenberg S, Meriggiola MC, Meuleman E, Mulders PF, Nieschlag E, Perheentupa A, Solomon A, Vaisala L, Wu FC, Zitzmann M. Male hormonal contraception: a double-blind, placebo-controlled study. J Clin Endocrinol Metab. 2008 Jul;93(7):2572-80. doi: 10.1210/jc.2008-0265. Epub 2008 Apr 15. PMID 18413423